CLINICAL TRIAL: NCT04879290
Title: Comparison of Two FiO2 (1 or 0.5) for Tracheal Extubation in Post-anesthesia Care Unit : a Monocentric Randomized Trial
Brief Title: Comparison of Two FiO2 (1 or 0.5) for Tracheal Extubation in Post-anesthesia Care Unit
Acronym: EXTUBO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-172
Record Dates: First submitted 2021-04-23; First posted 2021-05-10 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia; Atelectasis; Postoperative Complications; Hypoxemia; Hyperoxia
Keywords: Post-anesthesia care unit; Extubation
MeSH Terms: conditions — Pulmonary Atelectasis; Postoperative Complications; Hypoxia; Hyperoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group FiO2=1 (Active Comparator): FiO2 = 1 (100%) 10mn before emergence of general anesthesia
  Interventions: Other: FiO2 1
- Intervention Group FiO2 0.5 (Experimental): Fi02 = 0.5 (50%) 10mn before emergence of general anesthesia
  Interventions: Other: FiO2 0.5

INTERVENTIONS:
Other: FiO2 0.5 — Ten minutes before emergence from general anesthesia, the amount of oxygen delivered from the mechanical ventilator called fractional inspired oxygen (FiO2) is set to 0.5 (50%)
  Arms: Intervention Group FiO2 0.5
Other: FiO2 1 — Ten minutes before emergence from general anesthesia, the amount of oxygen delivered from the mechanical ventilator called fractional inspired oxygen (FiO2) is set to 1 (100%)
  Arms: Control Group FiO2=1

SUMMARY:
The purpose of the study is to assess the optimal fraction of inspired oxygen (0.5 or 1) for extubation or removal of a supraglottic airway device after general anesthesia.

DETAILED DESCRIPTION:
During pre-anesthesia visit, eligible patients receive oral and written information of the study and potential risks.

In the operating room all patients giving a written informed consent will undergo at the end of surgery a screening to determine eligibility for study entry.

Before emergence from general anesthesia, patients who meet the eligibility requirements will be randomized in a open label manner to receive a 0.5 or 1 FiO2.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia, with invasive mechanical ventilation including an airway device (supraglottic airway device or tracheal tube) at their arrival in PACU.
* ASA physical status classification 1, 2, or 3 stabilized.
* Surgery performed in emergency operating room department including vascular, digestive, urological and minor trauma surgery or surgery performed in head and neck anesthesia pole block including anterior cervical spine, lumbar disc herniation, cranioplasty, nerve stimulator, vertebroplasty, narrow lumbar canal, simple arthrodesis (less than or equal to two stages), otological, ophthalmological and skin surgery.

Exclusion Criteria:

* Per-operative hemodynamic instability.
* Patients with a BMI greater than 35.
* Patients classified as difficult to intubate and / or ventilate.
* Heavy surgeries (operating time greater than 4 hours).
* Patient requiring postoperative non invasive mechanical ventilation
* Patients with diagnosed COPD
* SPO2 in room air < 96% before the intervention.
* Any patient under guardianship.
* Pre-operative and / or intra-operative morphine intake.
* Surgical management of the upper airways (ex : tonsillectomy)
* Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Decrease of oxygen saturation | Duration of stay in post-anesthesia care unit, approximately one hour
  Proportions of patients that present a decrease of 4 points of peripheral capillary oxygen saturation (SpO2) measured with pulse oximetry after extubation compared to their baseline room air SpO2

SECONDARY OUTCOMES:
Duration of emergence | Up to one hour
  Elapsed Time between cessation of sedation and extubation (minutes)
Primary Outcome Timing | Up to one hour
  Elapsed time between extubation and decrease of oxygen saturation (minutes)
Number of risk factors | One hour
  Number of factors associated with episodes of hypoxemia : bronchospasm, bronchial congestion (profuse secretions with the need to aspirate the patient several times), loss of upper airway muscle tonus (fall of the tongue).
Majored decrease of oxygen saturation | One hour
  Proportions of patients that present a decrease of 6 points of SpO2 after extubation compared to their baseline room air SpO2
Corrective measures | One hour
  Number of corrective measures (method and oxygen supply equipment used) after hypoxemia and proportion of success.
PACU length of stay | One hour
  Length of stay in post-anesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Dr KAMGA TOTOUOM, MD, Principal Investigator — Anesthesiologist; Pr HANOUZ, PhD, Study Director — Anesthesiologist; Dr BOUTROS, MD, Principal Investigator — Anesthesiologist
Locations (1):
- University Hospital, Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No